CLINICAL TRIAL: NCT05262699
Title: SFB TRR 169/A3 (2.FP) Crossmodal Learning in Health and Neurological Disease: Neurocomputational Representation and Therapeutic Application (Task 2-1)
Brief Title: Crossmodal Learning in Therapeutic Processes (Task 2-1)
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Unability to include participants during Covid pandemic
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: German Research Foundation (Other); National Natural Science Foundation of China (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SFB TRR 169/A3 (2-1)
Record Dates: First submitted 2022-02-05; First posted 2022-03-02 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Stroke
Keywords: Vibro-tactile stimulation; Neurorehabilitation; Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Assessment, motor training, data analyzes, and group allocation are done by different persons. Participants as well as the assessor, the trainer and the investigator are blinded to the group allocation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stimulation (Experimental): During motor training participants in the stimulation arm receive vibro-tactile feedback applied to their fingers when touching an object as measured by force-sensing resistors mounted to the fingertips.
  Interventions: Device: Vibro-tactile stimulation
- Control (Placebo Comparator): The control group receives the same motor training with the same derives (force-sensing resistors, vibro-tactile stimulators) mounted to the hands but receives no stimulation.
  Interventions: Other: Placebo Control

INTERVENTIONS:
Device: Vibro-tactile stimulation — Vibro-tactile stimulation will be administered to the fingers of the participants via C3 tactors (diameter: 2.03 cm, height: 0.64 cm, operating frequency: 180-320 Hz, see https://www.eaiinfo.com/tactor-info/). Vibro-tactile stimulation will be triggered by force-sensing resistors (TEA CAPTIV T-SENS FSR, see https://www.teaergo.com/products/tea-captiv-t-sens-fsr/).
  Arms: Stimulation
Other: Placebo Control — Devices mounted, no stimulation
  Arms: Control

SUMMARY:
Interventional study of the effects of vibro-tactile feedback on behavioral deficits and learning during motor training in patients with stroke.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic stroke according to ICD 10 I61-I69
* Deficit still existing (Rankin score of at least 1 at inclusion)
* Age >= 18, <=80
* Existing declaration of consent

Exclusion Criteria:

* Pregnancy
* Lacking capacity for consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2021-04-14 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Action Research Arm Test (ARAT) | One day before (baseline) and one day after seven days of motor training
  The Action Research Arm Test (ARAT) is a 19 item observational measure to assess upper extremity performance (coordination, dexterity and functioning). Items comprising the ARAT are categorized into four subscales (grasp, grip, pinch and gross movement) and arranged in order of decreasing difficulty, with the most difficult task examined first, followed by the least difficult task. Task performance is rated on a 4-point scale, ranging from 0 (no movement) to 3 (movement performed normally). Scores may range from 0-57 points, with higher points indicating better performance.
Change from baseline in Nine-hole peg Test (NHPT) | One day before (baseline) and one day after seven days of motor training
  A timed measure of fine manual dexterity where the patient is instructed to first take nine pegs out of a container and place them afterwards back into the empty holes of the container as quickly as possible.

SECONDARY OUTCOMES:
Change from baseline in Fugl-Meyer Assessment for upper extremity (FMA-UE) | One day before (baseline) and one day after seven days of motor training
  The section motor function of upper limb is one of five domains, a three-point scale is used for rating performance as 0=cannot perform, 1=performs partially and 2=performs fully, max. possible score: 66 points.
Change from baseline in Stroke Impact Scale (SIS) | One day before (baseline) and one day after seven days of motor training
  Measurement of subjective stroke-specific health status, 64 items in eight domains, domain scores range between 0-100, with higher scores represent better health status.
Change from baseline in National Institutes of Health Stroke Scale (NIHSS) | One day before (baseline) and one day after seven days of motor training
  The National Institutes of Health Stroke Scale, NIHSS, is a score system to quantify the impairment caused by a stroke. The sum of the values from the investigations results in a maximum of 42 points. The higher the score, the more extensive the stroke.
Change from baseline in Modified Rankin Scale (mRS) | One day before (baseline) and one day after seven days of motor training
  The modified Rankin scale (MRS) is a standardized measure that describes the extent of disability after a stroke. It ranges from 0 (no symptoms) to 6 (death due to stroke).

CONTACTS AND LOCATIONS:
Locations (1):
- Universitätsklinikum Hamburg-Eppendorf, Neurologie, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: Yes
Data sharing is planned after main publication of results.
Supporting Information: Study Protocol
Time Frame: Within 24 months after main publication.
Access Criteria: Personal login into UKE data repository.